CLINICAL TRIAL: NCT05887817
Title: Effects of Finerenone on Vascular Stiffness and Cardiorenal Biomarkers in Type 2 Diabetes and Chronic Kidney Disease (FIVE-STAR)
Brief Title: Effects of Finerenone on Vascular Stiffness and Cardiorenal Biomarkers in T2D and CKD (FIVE-STAR)
Acronym: FIVE-STAR
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Saga University (Other)
Responsible Party: Principal Investigator, Koichi Node, Professor, Saga University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00002
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes; Chronic Kidney Diseases
Keywords: Finerenone; Vascular Stiffness; Biomarker
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — finerenone

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Finerenone (Experimental): Kerendia® tablets
  Interventions: Drug: Finerenone
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finerenone — Study participants will be instructed to take either finerenone or placebo orally once daily (preferably at approximately the same time every during the morning). For study participants with baseline eGFR less than 60mL/min/1.73 m2, the starting dose will be 10mg/day of finerenone (equivalent to 10mg/day in the placebo group), followed by 20 mg/day (equivalent to 20mg/day in the placebo group) approximately 4 weeks after the first dose, in accordance with the latest package insert. The dose should be increased to 20mg/day (equivalent to 20mg/day in the placebo group) in principle after 4 weeks from the start of the first dose, in accordance with the latest package insert. Study participants with a baseline eGFR of 60 mL/min/1.73m2 or higher will receive 20mg/day of finerenone (equivalent to 20mg/day in the placebo group) as the starting dose.
  Other Names: Kerendia
  Arms: Finerenone
Drug: Placebo — Study participants will be instructed to take either finerenone or placebo orally once daily (preferably at approximately the same time every during the morning). For study participants with baseline eGFR less than 60mL/min/1.73 m2, the starting dose will be 10mg/day of finerenone (equivalent to 10mg/day in the placebo group), followed by 20 mg/day (equivalent to 20mg/day in the placebo group) approximately 4 weeks after the first dose, in accordance with the latest package insert. The dose should be increased to 20mg/day (equivalent to 20mg/day in the placebo group) in principle after 4 weeks from the start of the first dose, in accordance with the latest package insert. Study participants with a baseline eGFR of 60 mL/min/1.73m2 or higher will receive 20mg/day of finerenone (equivalent to 20mg/day in the placebo group) as the starting dose.
  Arms: Placebo

SUMMARY:
To evaluate the effects of finerenone on vascular stiffness and cardiorenal biomarkers in patients with type 2 diabetes and chronic kidney disease.

DETAILED DESCRIPTION:
Finerenone is a novel non-steroidal selective mineralocorticoid receptor antagonist (MRA), characterized by a higher selectivity and affinity for mineralocorticoid receptors than conventional steroidal MRA. In the international phase III trials (FIDELIO-DKD and FIGARO-DKD), finerenone reduced the risk of progression of nephropathy and cardiovascular events in chronic kidney disease (CKD) patients with type 2 diabetes (T2D) who had been on standard treatment for CKD and T2D. However, the possible mechanistic insights into clinical benefits of finerenone in that patient population are currently very limited. To address them, in this investigator-initiated, multicenter, placebo-controlled, randomized trial (FIVE-STAR), the investigators seek to assess the effects of finerenone on vascular stiffness and cardiorenal biomarkers in patients with T2D and CKD.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given their written consent to participate in this study
* Patients who are 20 years of age or older at the time of consent (regardless of gender)
* Patients with type 2 diabetes mellitus
* Patients with chronic kidney disease who meet both of the following criteria; i) eGFR greater than 25 mL/min/1.73 m2 and less than 90 mL/min/1.73 m2, ii) UACR greater than 30 mg/g.cr. and less than 3500 mg/g.cr.
* Patients who have not changed their medications for type 2 diabetes and chronic kidney disease in the past 4 weeks prior to obtaining consent

Exclusion Criteria:

* Patients who are currently taking or have taken MRAs containing finerenone in the past 4 weeks prior to obtaining consent.
* Patients with a history of hypersensitivity to finerenone
* Patients with HbA1c greater than 10%.
* Patients with a serum potassium level of 4.9 mEq/L or higher
* Patients with NYHA class II-IV HFrEF (LVEF <35%)
* Patients with poorly controlled hypertension (e.g., systolic BP >170 mmHg, diastolic BP >110 mmHg, or hypertensive emergencies)
* Patients with a history of ischemic stroke, acute coronary syndrome, cardiovascular surgery or percutaneous intervention, or hospitalization for worsening heart or renal failure in the past 8 weeks prior to obtaining consent
* Patients with a preplanned surgical or percutaneous intervention for coronary artery reconstruction or other cardiovascular disease during the individual observation period.
* Patients with a preplanned treatment such as electrical cardioversion, cardiac resynchronization therapy or pacemaker implantation during the individual observation period.
* Patients with preplanned dialysis or kidney transplantation during the individual observation period.
* Patients with severe hepatic dysfunction (Child-Pugh Class C)
* Patients receiving itraconazole, ritonavir-containing products, atazanavir, darunavir, fosamprenavir, cobicistat-containing products, or clarithromycin, or ensitrelvir
* Patients with Addison's disease
* Patients with active infectious diseases
* Pregnant, possibly pregnant, or lactating patients
* Other patients deemed inappropriate for this study by the principal investigator or subinvestigators (e.g., patients with renal artery stenosis, one kidney, or active malignancy).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in CAVI | 24 weeks
  Change in CAVI at 24 weeks after initiation of protocol treatment compared to baseline

SECONDARY OUTCOMES:
Change in UACR | 12 weeks, 24 weeks
  Proportional changes in geometric mean of UACR at 12 and 24 weeks post-protocol treatment compared to baseline (key secondary endpoint)
Change in pentosidine | 24 weeks
  Proportional changes in geometric mean of pentosidine at 24 weeks post-protocol treatment compared to baseline
Change in urinary type IV collagen | 24 weeks
  Proportional changes in geometric mean of urinary type IV collagen at 24 weeks post-protocol treatment compared to baseline
Change in urinary alpha1-MG | 24 weeks
  Proportional changes in geometric mean of urinary alpha1-MG at 24 weeks post-protocol treatment compared to baseline
Change in urinary beta2-MG | 24 weeks
  Proportional changes in geometric mean of urinary beta2-MG at 24 weeks post-protocol treatment compared to baseline
Change in urinary NGAL | 24 weeks
  Proportional changes in geometric mean of urinary NGAL at 24 weeks post-protocol treatment compared to baseline
Change in urinary NAG | 24 weeks
  Proportional changes in geometric mean of urinary NAG at 24 weeks post-protocol treatment compared to baseline
Change in urinary L-FABP | 24 weeks
  Proportional changes in geometric mean of urinary L-FABP at 24 weeks post-protocol treatment compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Koichi Node, MD, PhD, Principal Investigator — Saga University Hospital
Locations (1):
- Saga University Hospital, Saga, Japan

REFERENCES:
- [Derived] Tanaka A, Shibata H, Imai T, Yoshida H, Miyazono M, Takahashi N, Fukuda D, Okada Y, Teragawa H, Suwa S, Kida K, Moroi M, Taguchi I, Toyoda S, Shimabukuro M, Tanabe K, Tanaka K, Nangaku M, Node K; FIVE-STAR trial investigators. Rationale and design of an investigator-initiated, multicenter, prospective, placebo-controlled, double-blind, randomized trial to evaluate the effects of finerenone on vascular stiffness and cardiorenal biomarkers in type 2 diabetes and chronic kidney disease (FIVE-STAR). Cardiovasc Diabetol. 2023 Jul 31;22(1):194. doi: 10.1186/s12933-023-01928-y. PMID 37525257